CLINICAL TRIAL: NCT04001712
Title: Effect of Early Use of Caffeine Citrate in Preterm Neonates Needing Respiratory Support.
Brief Title: Effect of Early Use of Caffeine Citrate in Preterm Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: early caffeine in preterm
Record Dates: First submitted 2019-06-22; First posted 2019-06-28 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Preterm Birth
Keywords: early caffeine preterm
MeSH Terms: conditions — Premature Birth | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: randomized controlled phase 3 clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early caffeine citrate group (Experimental): preterm neonates who require respiratory support either nasal canula, continuous positive airway pressure (CPAP) or mechanical ventilation.were given caffeine citrate upon start of the respiratory support Caffeine citrate was given at a loading dose of 10 mg/kg and with a daily maintenance dose of 5 mg/kg until the patient was off respiratory support
  Interventions: Drug: Caffeine Citrate
- late caffeine citrate group (Active Comparator): preterm neonates who require respiratory support either nasal canula, continuous positive airway pressure (CPAP) or mechanical ventilation.were given caffeine citrate 6 hours before weaning of respiratory support
  Interventions: Drug: Caffeine Citrate

INTERVENTIONS:
Drug: Caffeine Citrate — caffeine citrate is given early to preterm neonates in need of respiratory support

SUMMARY:
This work is designed to study the effect of the early use of caffeine citrate in preterm neonates who need respiratory support on morbidity and short term neonatal outcome.

DETAILED DESCRIPTION:
Caffeine citrate is one of the most widely used drugs in neonatal intensive care units. It is a respiratory stimulant which has well established therapeutic effects in apnea and facilitation of extubation. Caffeine is an adenosine antagonist ; it blocks selectively A2 receptors and non selective blocks A1 receptors. Its effects include improved lung compliance, minute ventilation, respiratory muscle contractility, increased sensitivity to carbon dioxide, enhanced catecholamine activity and decreased airway resistance

Early caffeine therapy was associated with a shorter duration of respiratory support and reduction in bronchopulmonary dysplasia , cerebral palsy, patent ductus arteriosis ligation, intracranial hemorrhage, apnea and death

Despite its widespread use, information regarding optimal time to initiate therapy and appropriate time to discontinue therapy is limited. Recent studies have indicated that early initiation of caffeine therapy is associated with improved neonatal outcomes

Little is known about the early use of caffeine citrate in preterm neonates. The investigators aim to explore the effectiveness of its very early use in reducing the duration of respiratory support.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm neonates ≤ 33 weeks gestational age.
2. Preterm neonates who need respiratory support (either nasal canula, continuous positive airway pressure (CPAP) or mechanical ventilation).

Exclusion Criteria:

1. Neonate>33 wks gestational age.
2. Neonates on room air.
3. Neonates with major congenital or cardiac anomalies

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
duration of respiratory support in preterm neonates receiving early caffeine citrate | throughout admission in neonatal intensive care unit average of 4 weeks (from the beginning of hospital admission till discharge) average of
  preterm neonates of gestational age 33 weeks or less needing any respiratory support (CPAP , mechanical ventilation....)were given caffeine citrate at the start of the support. duration of the support was compared to the duration of respiratory support in the other arm that includes preterm neonates of gestational age 33 weeks or less needing any respiratory support and receiving caffeine citrate 6 hours before weaning only.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem El Sayed, Study Chair — Ain Shams University; Sameh Amer, Study Chair — Medical Military Academy; Hisham Awad, Study Director — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Lista G, Fabbri L, Polackova R, Kiechl-Kohlendorfer U, Papagaroufalis K, Saenz P, Ferrari F, Lasagna G, Carnielli VP; Peyona(R) PASS Group. The Real-World Routine Use of Caffeine Citrate in Preterm Infants: A European Postauthorization Safety Study. Neonatology. 2016;109(3):221-7. doi: 10.1159/000442813. Epub 2016 Jan 28. PMID 26820884
- [Background] Lodha A, Seshia M, McMillan DD, Barrington K, Yang J, Lee SK, Shah PS; Canadian Neonatal Network. Association of early caffeine administration and neonatal outcomes in very preterm neonates. JAMA Pediatr. 2015 Jan;169(1):33-8. doi: 10.1001/jamapediatrics.2014.2223. PMID 25402629
- [Background] Rivera-Oliver M, Diaz-Rios M. Using caffeine and other adenosine receptor antagonists and agonists as therapeutic tools against neurodegenerative diseases: a review. Life Sci. 2014 Apr 17;101(1-2):1-9. doi: 10.1016/j.lfs.2014.01.083. Epub 2014 Feb 13. PMID 24530739